CLINICAL TRIAL: NCT03857607
Title: Natural History of ATP1A3-related Disease: a Deep Phenotyping-genotyping Project
Brief Title: Natural History Study of ATP1A3-related Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17NC04
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: ATP1A3-related Disease; Alternating Hemiplegia of Childhood; Rapid Onset Dystonia Parkinsonism; CAPOS
MeSH Terms: conditions — Alternating hemiplegia of childhood; Dystonia 12; CAPOS syndrome | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Whole exome sequencing — Whole exome sequencing will be used to identify causative genes in ATP1A3 mutation negative patients, to confirm causality in ambiguous phenotypes and to identify modifier genes.

SUMMARY:
An observational study aiming to study the natural history of a UK-wide patient cohort with ATP1A3-related disease.

DETAILED DESCRIPTION:
Alternating hemiplegia of childhood (AHC) is a rare very disabling neurodevelopmental syndrome caused by mutations in the gene ATP1A3. AHC is characterized by paroxysmal events including attacks of hemiplegia (weakness), dystonia (painful stiffening), oculomotor abnormalities and epileptic seizures. As the condition progresses permanent neurological symptoms, including unsteadiness and learning problems, emerge. Mutations in ATP1A3 also cause other related syndromes: rapid-onset dystonia-parkinsonism (RDP), less severe and usually presenting in adulthood, as well as cerebellar ataxia, areflexia, pes cavus, optic atrophy, and sensorineural hearing loss (CAPOS) syndrome, a severe syndrome of early childhood.

Currently therapeutic options are very limited aiming at symptomatic relief with limited success. As ATP1A3-related syndromes are very rare diseases, with an estimated prevalence of about 1/1000000, randomised clinical trials of available therapies are not possible due to lack of a large enough patient cohort. However, the revolution in genetic diagnostics has made the identification of these patients and the correlation between their phenotypes possible. At the same time further novel technologies in neuromonitoring and neuroimaging, as well as videography and sleep monitoring have become available that could help us further examine and understand the underlying mechanisms especially of the paroxysmal episodes that characterise all ATP1A3-related syndromes. The investigators believe that based on these scientific advances they will be able to recruit a UK-wide patient cohort to conduct an in depth study of the progression of this disease.

This is particularly relevant at the moment as rapid progress in genetic therapies and other novel therapeutics makes the availability of new treatment options in the near future a realistic prospect and, even though we will most probably still not be able to identify a large enough cohort for randomised clinical trials, our natural history study will act as a much needed benchmark to which the success of novel treatments can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults of any age carrying a mutation in the ATP1A3-gene.
* Children and adults of any age matching an ATP1A3-related disease phenotype without a mutation in the gene.
* Written informed consent given by patient and/or parent/guardian.

Exclusion Criteria:

• Patients with a phenotype not fitting ATP1A3-related disease and no mutation in the ATP1A3 gene.

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: UK-wide cohort of patients carrying an ATP1A3-mutation or diagnosed with a phenotype associated with ATP1A3-related disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Cross, PhD, Principal Investigator — UCL Institute of Child Health
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No